CLINICAL TRIAL: NCT01854255
Title: Feasibility, Efficacy and Safety of Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) With Cisplatin and Doxorubicin in Patients With Gastric Cancer and Peritoneal Carcinomatosis: an Open-label, Single-arm, Phase II Clinical Trial
Brief Title: Intraperitoneal Aerosol Chemotherapy in Gastric Cancer
Acronym: PIPAC-GA01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Clemens Tempfer, Clemens Tempfer, MD, MBA, Ruhr University of Bochum
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIPAC-GA01
Record Dates: First submitted 2013-05-12; First posted 2013-05-15 (Estimated); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Gastric Cancer
Keywords: Gastric; Cancer; Chemotherapy; Intraperitoneal
MeSH Terms: conditions — Stomach Neoplasms; Neoplasms | interventions — Doxorubicin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intraperitoneal Chemotherapy (Experimental): Patients will receive doxorubicin 1.5 mg/m2 body surface in 50 ml NaCl 0,9% and cisplatin 7.5 mg/m2 in 50 ml NaCl 0,9% q 4-6 weeks, applied intraperitoneally as pressurized aerosol chemotherapy. Duration of treatment will be 3 single doses in 6 weeks intervals, thus the duration of treatment is 18 weeks.
  Interventions: Drug: doxorubicin and cisplatin

INTERVENTIONS:
Drug: doxorubicin and cisplatin — doxorubicin and cisplatin as intraperitoneal chemotherapy
  Other Names: doxorubicin 50 HEXAL®; cisplatin 10 HEXAL®

SUMMARY:
A prospective series of patients with recurrent gastric cancer will be treated with three cycles of chemotherapy (doxorubicin and cisplatin) instilled into the abdominal cavity in the form of an aerosol under pressure via laparoscopy. The efficacy of this treatment will be assessed by computed tomography, tumor marker studies, and survival. Also, the safety of the procedure will be assessed.

DETAILED DESCRIPTION:
Objectives: To evaluate the safety and efficacy in terms of the clinical benefit rate (CBR) of PIPAC in peritoneal carcinomatosis (PC) from gastric cancer (GC) Study design: Single center, open label, non-randomized, single-arm, repeated single dose study to explore the efficacy, safety, and CBR of doxorubicin and cisplatin when given as a pressurized intraperitoneal aerosol chemotherapy (PIPAC) to patients with advanced gastric cancer and peritoneal carcinomatosis.

Target subject population:Patients with GC and PC with disease progression after at least one line of previous i.v. chemotherapy.

Investigational product, dosage and mode of administration Doxorubicin 1.5 mg/m2 body surface in 50 ml NaCl 0,9% and Cisplatin 7.5 mg/m2 in 50 ml NaCl 0,9% q 4-6 weeks, applied intraperitoneally as PIPAC.

Duration of treatment: 3 single doses in 6 weeks intervals, duration of treatment is 18 weeks

Outcome variables:

1.1 Primary outcome variable • Clinical Benefit Rate (CBR) according to Response Evaluation Criteria In Solid Tumors (RECIST) criteria (version 1.1) after 3 cycles of PIPAC with cisplatin and doxorubicin.

1.2 Secondary outcome variables

* The observed survival (OS)
* The median time to progression (TTP) according to RECIST criteria after three cycles of PIPAC with cisplatin and doxorubicin
* The Peritoneal Carcinomatosis Index (PCI) before and after therapy
* The degree of histological regression assessed by pathological review
* Apoptosis as assessed by immunohistochemical analysis
* The difference in ascites volume before and after the first, second, and third PIPAC application 1.3 Patient reported outcomes (PROs)
* European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ-C30, German version ) 1.4 Safety
* Safety and tolerability will be assessed by collection of adverse events, according to the Common Terminology Criteria for Adverse Events (CTCAE) including physical examination results, laboratory assessments (chemistry and hematology).

1.5 Biological monitoring

• Basic research investigating expression of genes associated with drug resistance.

ELIGIBILITY:
Inclusion Criteria:

* age above 18 years
* written, informed consent
* presence of peritoneal carcinomatosis

Exclusion Criteria:

* language barrier
* parenchymal metastases
* unability to undergo laparoscopy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-11; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Clinical Benefit Rate | within 3 months after treatment completion
  Clinical Benefit Rate according to RECIST criteria after 3 cycles of PIPAC with cisplatin and doxorubicin.

SECONDARY OUTCOMES:
Observed Survival | During treatment and follow-up of 1 year
  Survival will be assessed by direct observation during treatment and by follow-up investigation for 1 year after completion of the study

OTHER OUTCOMES:
median time ot progression | during treatment and follow-up of 1 year
  Time to progression according to RECIST criteria during treatment and during follow-up of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marc A Reymond, MD, Principal Investigator — Ruhr University of Bochum
Locations (1):
- Ruhr University of Bochum, Herne, North Rhine-Westphalia, Germany

REFERENCES:
- [Result] Struller F, Horvath P, Solass W, Weinreich FJ, Strumberg D, Kokkalis MK, Fischer I, Meisner C, Konigsrainer A, Reymond MA. Pressurized intraperitoneal aerosol chemotherapy with low-dose cisplatin and doxorubicin (PIPAC C/D) in patients with gastric cancer and peritoneal metastasis: a phase II study. Ther Adv Med Oncol. 2019 May 13;11:1758835919846402. doi: 10.1177/1758835919846402. eCollection 2019. PMID 31205501